CLINICAL TRIAL: NCT05843838
Title: The Effect of Intraoperative Hypotension on Postoperative Cognitive Functions in Cesarean Section Operations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E2-23-3719
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: cesarean section; postoperative cognitive dysfunction; hypotension
MeSH Terms: conditions — Postoperative Cognitive Complications; Hypotension | interventions — Cesarean Section; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypotensive group (Experimental): Patients who are hypotensive (even once) and need ephedrine under spinal anesthesia with routine doses of heavy bupivacaine (Hypotension, Mean Arterial Pressure<65 mmHg, or Systolic arterial pressure < 30% will be considered an initial value.)
  Interventions: Procedure: Hypotension during spinal anesthesia for cesarean section; Diagnostic Test: Mini-mental test; Procedure: Spinal anesthesia; Diagnostic Test: The Bromage scale; Drug: Heavy Bupivacaine for spinal anesthesia
- Normotensive group (Placebo Comparator): Patients who are not hypotensive under spinal anesthesia with routine doses of heavy bupivacaine
  Interventions: Diagnostic Test: Mini-mental test; Procedure: Spinal anesthesia; Diagnostic Test: The Bromage scale; Drug: Heavy Bupivacaine for spinal anesthesia

INTERVENTIONS:
Procedure: Hypotension during spinal anesthesia for cesarean section — Hypotension, Mean Arterial Pressure<65 mmHg, or Systolic arterial pressure < 30% will be considered an initial value
  Arms: Hypotensive group
Diagnostic Test: Mini-mental test — A Mini-Mental State test is a set of questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory).
  At the end of the research, the mental test scores of the two groups will be compared and the effect of hypotension will be evaluated.
Procedure: Spinal anesthesia — It is a neuraxial anesthesia technique in which local anesthetic is placed directly in the intrathecal space. Spinal anesthesia will be applied to both groups with heavy bupivacaine in usual doses.
Diagnostic Test: The Bromage scale — The Bromage scale is the accepted tool for motor block examination. The classification of these scores
  1. complete block: unable to move feet or knees
  2. almost complete: able to move feet only
  3. partial: just able to flex knees; free movement of feet
  4. no block: full movement of knees and feet
Drug: Heavy Bupivacaine for spinal anesthesia — Routine clinical heavy bupivacaine doses

SUMMARY:
The aim of the study is to see whether the hypotension that develops during spinal anesthesia in cesarean section patients causes a decrease in the postoperative cognitive functions of the patient. If the results show a decrease in functions due to the effect of hypotension, it will be necessary to carry out aggressive prevention/treatment of hypotension in cesarean section patients.

DETAILED DESCRIPTION:
A total of 150 female patients (75 in each group) between the ages of 18-40 who will undergo caesarean section with spinal anesthesia in the obstetric operating room of Ankara Bilkent City Hospital in ASA 2, 3rd categories will be included in the study.

Patients will be divided into two as hypotensive and non-hypotensive patients in spinal anesthesia with routine doses, and all patients will be given a mini mental test at preop and post op 1st hour. (Hypotension, MAP(mean artery pressure)<65 mmHg, or SAP(systemic arterial pressure) < 30% will be considered as an initial value.) Patients who are hypotensive and need ephedrine will be included in the hypotensive group, and patients without hypotension will be included in the normotensive group. Those with an initial mini mental test score below 24 will not be allowed to study. At the end of the research, the mental test scores of the two groups will be compared and the effect of hypotension will be evaluated.

The patient's name-surname, age, protocol number, indication for cesarean section, method of regional anesthesia applied, sensory block level, Bromage score, side effect follow-up, first ten minutes after the procedure, every two minutes, up to half an hour, and every fifteen minutes after thirty minutes, systolic artery pressure, diastolic artery pressure, average arterial pressure, pulse and ephedrine (if used) will be recorded.

Preoperative, Postoperative first hour Mini Mental Test Score will be administered and recorded

ELIGIBILITY:
Inclusion Criteria:

* Female patients between the ages of 18-40 in the ASA2, 3rd categories who will undergo cesarean section with spinal anesthesia who agree to participate in the study

Exclusion Criteria:

* Failure of the patient to accept
* The necessity of an additional intervention to the cesarean section
* Change of routine practices on a patient-by-patient basis with the occurrence of complications in the surgical process
* Presence of additional diseases
* Emergency cases, cases using intraoperative sedation
* Those who do not speak the language
* Those who have an initial Mini Mental Test score lower than 24

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative cognitive function related with hypotension in cesarean section | Preoperative (in 10 minutes before operation) to postoperative first hour.
  Postoperative cognitive dysfunction is defined as the decrease in postoperative 1st hour mini-mental test results compared to preoperative results.Higher scores of mini-mental test mean a better outcome.By comparing the difference between the preoperative and postoperative mini-mental test results of the patients in the two arms, It will be observed whether there is a cognitive function difference between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: esra uyar türkyılmaz, Principal Investigator — Ankara Bilkent City Hospital Ankara Turkey
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)